CLINICAL TRIAL: NCT03082144
Title: Involved-field Radiotherapy Combined With Concurrent Intrathecal-MTX Versus Intrathecal-Ara-C for Leptomeningeal Metastases From Solid Tumor: A Randomized Phase II Clinical Trial
Brief Title: Concurrent Involved-field Radiotherapy and Intrathecal Chemotherapy for Leptomeningeal Metastases From Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MVARTICLM
Record Dates: First submitted 2017-03-05; First posted 2017-03-17 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Cytarabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: RT-Intra-MTX (Active Comparator): Intrathecal chemotherapy: MTX 15 mg, plus dexamethasone 5 mg, via lumbar puncture,once per week, 4 weeks in total.
  Interventions: Drug: MTX; Radiation: Radiotherapy
- Group2: RT-Intra-Ara-C (Experimental): Intrathecal chemotherapy:Ara-C 50 mg, plus dexamethasone 5 mg, via lumbar puncture, once per week, 4 weeks in total.
  Interventions: Drug: Ara-C; Radiation: Radiotherapy

INTERVENTIONS:
Drug: MTX — MTX 15 mg,via lumbar puncture,once per week, 4 weeks in total
  Other Names: Intrathecal chemotherapy
  Arms: Group 1: RT-Intra-MTX
Drug: Ara-C — Ara-C 50mg,via lumbar puncture,once per week, 4 weeks in total
  Other Names: Intrathecal chemotherapy
  Arms: Group2: RT-Intra-Ara-C
Radiation: Radiotherapy — The sites of symptomatic disease, bulky disease observed on MRI, including the whole brain and basis cranii, 40 Gy in 20 fractions;and/or segment of spinal canal received 40-50 Gy in 20-25 fractions.

SUMMARY:
It has been proved that concurrent radiotherapy (RT) and intrathecal methotrexate (MTX) for leptomeningeal metastases (LM) from solid tumors with adverse prognostic factors showed great effectiveness and safety. Cytarabine(Ara-C) is another agent which is commonly used for intrathecal chemotherapy. The purpose of the study is to observe the effectiveness and safety of concurrent RT and intrathecal chemotherapy for LM from solid tumors. In addition, the effectiveness of these two types of agents (MTX and Ara-C) in the concurrent chemo-radiotherapy will be compared in this study. This is a randomized controlled, parallel group, and phase II clinical trial. The object of this study is newly diagnosis patients with leptomeningeal metastases from solid tumors, who will accept the treatment of involved-field RT combined with concurrent intrathecal-MTX or intrathecal-Ara-C, respectively. Major endpoint is clinical response rate. Secondary endpoints are time to progression,severe adverse events and overall survival.

DETAILED DESCRIPTION:
The patients were randomly divided into two groups, who will accept the treatment of involved-field RT combined with concurrent intrathecal-MTX or intrathecal-Ara-C, respectively. Concomitant regimen consisted of intrathecal chemotherapy (via lumbar puncture, MTX 15 mg, plus dexamethasone 5 mg, or Ara-C 50mg, plus dexamethasone 5 mg, once per week, 4 weeks in total) and RT. RT consisted of fractionated, conformal radiation given at a daily dose of 2 Gy. The planning volume consisted of sites of symptomatic disease, bulky disease observed on MRI, including the whole brain and basis cranii received 40 Gy in 20 fractions and/or segment of spinal canal received 40-50 Gy. The RANO proposal for response criteria of LM disease was used to assess the clinical response in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been definitely diagnosed as leptomeningeal metastasis according to cerebrospinal fluid cytology or neuroimaging, or patients who got the clinical diagnosis by combining with the history of cancer, clinical manifestation, cerebrospinal fluid examination, neuroimaging etc;
2. Patients who have been diagnosed as malignant solid tumor with definite pathologic type, excluding hematological malignancies (e.g., leukemia and lymphoma) or primary brain tumors;
3. No severe abnormal liver and kidney function; WBC≥2500/mm3, Plt≥60000/mm3;
4. No other severe chronic diseases;
5. No history of severe nervous system disease;
6. No severe dyscrasia;
7. Signed informed consent form.

Exclusion Criteria:

1. Patients with leptomeningeal metastasis from unknown primary tumor;
2. Patients who had received radiotherapy to the brain in the past 6 months;
3. Patients who had accepted systemic chemotherapy within one month before the treatment, or molecular targeted therapy less than 3 months;
4. Patients with poor compliance, or for other reasons, the researchers considered unsuitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical Response Rate (CRR) | The evaluation was performed once per week from the beginning of LM-related therapy, till 4 weeks later after concomitant therapy.
  The RANO proposal for response criteria of LM disease was used to assess the clinical response in this study.

SECONDARY OUTCOMES:
Incidence of severe adverse events (SAE) | At least 7 months after LM diagnosis or until death.
  Adverse events (AEs) were evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03). Events of grade 3-5 was defined as moderate and severe adverse events.
Overall survival(OS) | At least 7 months after LM diagnosis or until death.
  Survival time was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, Professor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Result] Pan Z, Yang G, He H, Zhao G, Yuan T, Li Y, Shi W, Gao P, Dong L, Li Y. Concurrent radiotherapy and intrathecal methotrexate for treating leptomeningeal metastasis from solid tumors with adverse prognostic factors: A prospective and single-arm study. Int J Cancer. 2016 Oct 15;139(8):1864-72. doi: 10.1002/ijc.30214. Epub 2016 Jun 30. PMID 27243238
- [Result] Pan Z, Yang G, Wang Y, He H, Pang X, Gao Y, Shi W, Li Y, Dong L, Song Y. Thinprep plus Papanicolaou stain method is more sensitive than cytospin-coupled Wright Giems stain method in cerebrospinal fluid cytology for diagnosis of leptomeningeal metastasis from solid tumors. PLoS One. 2015 Apr 7;10(4):e0122016. doi: 10.1371/journal.pone.0122016. eCollection 2015. PMID 25850010
- [Result] Pan Z, Yang G, Yuan T, Pang X, Wang Y, Qu L, Dong L. Leptomeningeal metastasis from hepatocellular carcinoma with other unusual metastases: a case report. BMC Cancer. 2014 Jun 3;14:399. doi: 10.1186/1471-2407-14-399. PMID 24893802
- [Result] Pan Z, Yang G, Wang Y, Yuan T, Gao Y, Dong L. Leptomeningeal metastases from a primary central nervous system melanoma: a case report and literature review. World J Surg Oncol. 2014 Aug 20;12:265. doi: 10.1186/1477-7819-12-265. PMID 25142885
- [Result] Mack F, Baumert BG, Schafer N, Hattingen E, Scheffler B, Herrlinger U, Glas M. Therapy of leptomeningeal metastasis in solid tumors. Cancer Treat Rev. 2016 Feb;43:83-91. doi: 10.1016/j.ctrv.2015.12.004. Epub 2015 Dec 24. PMID 26827696
- [Result] Grewal J, Saria MG, Kesari S. Novel approaches to treating leptomeningeal metastases. J Neurooncol. 2012 Jan;106(2):225-34. doi: 10.1007/s11060-011-0686-2. Epub 2011 Aug 28. PMID 21874597
- [Result] Chamberlain MC. Leptomeningeal metastasis. Curr Opin Oncol. 2010 Nov;22(6):627-35. doi: 10.1097/CCO.0b013e32833de986. PMID 20689429
- [Result] Chamberlain MC. Leptomeningeal metastasis. Curr Opin Neurol. 2009 Dec;22(6):665-74. doi: 10.1097/WCO.0b013e3283322a92. PMID 19738466
- [Result] Le Rhun E, Taillibert S, Chamberlain MC. Carcinomatous meningitis: Leptomeningeal metastases in solid tumors. Surg Neurol Int. 2013 May 2;4(Suppl 4):S265-88. doi: 10.4103/2152-7806.111304. Print 2013. PMID 23717798

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03082144/Prot_SAP_000.pdf